CLINICAL TRIAL: NCT02595255
Title: Antimüllerian Hormone as a Predictor of Future Infertility Risk in Prepubertal/Pubertal Cancer Patients
Brief Title: AMH as a Predictor of Infertility Risk in Children With Cancer (CHANCE)
Acronym: CHANCE
Status: Recruiting | Type: Observational
Sponsor: Erasme University Hospital (Other)
Collaborators: Queen Fabiola Children's University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CHANCE (CHildren, Amh, caNCEr)
Record Dates: First submitted 2015-11-02; First posted 2015-11-03 (Estimated); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Fertility Preservation; Lymphoma; Pediatrics Cancer; Gonadotropin-releasing Hormone Agonist
Keywords: chemotherapy/GnRH (gonadotropin-releasing hormone) analogues/lymphoma/children/fertility
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum for hormonal assessment
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- High risk: Conditioning therapy for bone marrow transplantation or pelvic irradiation. Fertility preservation is usually already proposed in this group of patients. No intervention.
  Interventions: Other: No intervention
- Moderate/low risk: Pathologies treated with chemotherapy regimen with moderate or low risk of inducing ovarian function insufficiency: AML (Acute myeloide leukemia), osteosarcoma, Ewing sarcoma, neuroblastoma, non-Hodgkin lymphoma, Hodgkin lymphoma, soft tissue sarcoma, ALL (acute lymphoblastic hormone), Wilms tumour, retinoblastoma.
  This is the study group we will compare with high risk and no risk patients. No intervention
  Interventions: Other: No intervention
- No risk: Patients with chronic benign diseases or malignancies who don't receive any chemotherapy or other gonadotoxic treatment.
  No intervention
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
While most of the children spontaneously recover menstruation or experienced normal puberty after chemotherapy, their ovarian reserve may be impaired by treatment inducing future infertility. Fertility preservation is currently proposed for selected prepubertal patients with a high risk of premature ovarian failure after treatment (mostly conditioning regimen for bone marrow transplantation). For patients with low or moderate risks, counselling is very difficult and no fertility preservation procedure is usually proposed for these patients as no marker of the ovarian reserve has been validated in this young population to assess the individual risk.

The primary objective of the study is to prevent long-term treatment-related infertility by detecting the young patients who normally progressed to menarche but have a reduced ovarian reserve. These patients may benefit from particular follow-up and fertility preservation procedure.

DETAILED DESCRIPTION:
In this clinical trial, we will prospectively evaluate the AMH (Antimüllerian Hormone) level before and after treatment (up to 18 years old) in a large cohort of pre- and post-pubertal children treated for cancer. The children enrolled are young patients between 3 and 14 year old who are newly diagnosed with cancer or benign diseases treated by chemotherapy and/or pelvic irradiation. They belong to one of these 3 groups (modified from Wallace et al, 2005):

* High risk
* Moderate/Low risk
* No risk (control group)

Primary endpoint:

Evaluate AMH as a potential biomarker of ovarian reserve in prepubertal/pubertal girl treated by chemotherapy (classified according to the AAD(Alkylating Agent Dose) score)

Secondary endpoints:

* Evaluate the association between the post-treatment ovarian reserve and the AMH pretreatment values in patients considered as moderate or low risk.
* Identify new patients group who may benefit from fertility preservation
* Compare the gonadotoxicity of chemotherapy regimen according to the pubertal status.
* Study the relation between the AMH levels and the pubertal age, menstruation cycle regularity, hormonal levels (FSH (follicle stimulating hormone), œstradiol, and testosterone) and bone age.

Different parameters will be assessed at inclusion, end of the treatment and during the follow-up (every year during the first 3 years and then every 2 years until the end of the study) Oncological outcome The patients will be followed up for progression and survival as per standard local practice.

Ovarian reserve and function:

Ovarian reserve will be evaluated based on hormonal dosages at different times of the study: FSH, AMH, estradiol, testosterone and LH (luteinizing hormone). Menstrual function will be evaluated by collecting information of the pubertal status (spontaneous or induced puberty) and menstrual cycle characteristics

Puberty evaluation:

All children will have an evaluation of the TANNER pubertal stage at 9 years of age (or later if > 9 years old at the time of inclusion) and once a year until the end of puberty (when patients reach Tanner stage 5). An X-ray of the left hand and wrist will be carried out for bone age evaluation at 9-11 and 13 years old.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 3 to 14 year old included - Belong to one of these 3 groups (modified from Wallace et al, 2005):

  * High risk : Conditioning therapy for bone marrow transplantation or pelvic irradiation
  * Moderate/Low risk : Pathologies treated with chemotherapy regimen with moderate or low risk of inducing ovarian function insufficiency: AML, osteosarcoma, Ewing sarcoma, neuroblastoma, non-Hodgkin lymphoma, Hodgkin lymphoma, soft tissue sarcoma, ALL, Wilms tumour, retinoblastoma.
  * No risk (control group) : patients with chronic benign diseases or malignancies who don't receive any chemotherapy or other gonadotoxic treatment.

Exclusion Criteria:

* CNS (central nervous system) irradiation, cerebral tumour
* Current or previous ovarian disease/surgery
* Familial history of premature ovarian failure (no iatrogenic or surgical origins)
* Previous known severe chronic disease potentially affecting normal growth or puberty (diseases inducing malnutrition, anorexia, genetic/congenital disorders as Turner, Kallman, BPES(Blepharophimosis, ptosis, and epicanthus inversus syndrome) syndromes, uncontrolled severe diabetes, Cushing Syndrome, auto-immune diseases, cystic fibrosis, severe renal dysfunction)
* Genetic/congenital disorders inducing mental retardation

Ages: 3 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Study Population: The population for this trial is patients between 3 and 14 year old newly diagnosed with cancer or benign diseases treated by chemotherapy and/or pelvic irradiation with high or moderate risk of inducing premature ovarian insufficiency. The "no risk" group includes patients with chronic benign diseases (as pneumology or gastroenterology diseases, congenital hypothyroidism, growth hormone deficiency or RCIU…) or malignancies who will not receive any chemotherapy or other gonadotoxic treatment.
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
AMH marker | screening, 1 year after screening, every year during the first 3 year of follow-up, every 2 years until 18 year old
  Blood test collection for serum storage. AMH values will be compared in the different groups and correlated with the cumulative doses of alkylating agents

SECONDARY OUTCOMES:
Premature ovarian failure (POF) | screening, 1 year after screening, every year during the first 3 year of follow-up, every 2 years until 18 year old
  Blood test collection for serum storage. FSH, E2 and AMH measurement and pubertal status. POF rate will be compared between groups
Ovarian reserve | screening, 1 year after screening, every year during the first 3 year of follow-up, every 2 years until 18 year old
  relation between the AMH levels, pubertal age, menstruation cycle regularity, hormonal levels (FSH, œstradiol, and testosterone at 16 year old) and bone age

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Demeestere, PhD, Study Director — Erasme ULB- Belgium; Alina Ferster, Principal Investigator — Queen Fabiola children's university hospital- Belgium; Christine Decanter, Principal Investigator — CHRU Lille, France
Locations (10):
- Belgium (7):
  - Centre Hospitalier Chrétien (CHC)- Clinique de l'espérance, Montegnée, Liège
  - Universitair Ziekenhuis Antwerpen, Antwerp
  - Hôpital Universitaire Reine Fabiola (HUDERF), Brussels
  - Universitair Ziekenhuis Brussels, Brussels
  - UZ-Gent, Ghent
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Régional (CHR)-Citadelle, Liège
- France (3):
  - Centre Oscar Lambret, Lille
  - CHRU Lille-Hôpital Jeanne de Flandre, Lille
  - Hôpital Robert Debré, Paris

REFERENCES:
- [Background] Brougham MF, Crofton PM, Johnson EJ, Evans N, Anderson RA, Wallace WH. Anti-Mullerian hormone is a marker of gonadotoxicity in pre- and postpubertal girls treated for cancer: a prospective study. J Clin Endocrinol Metab. 2012 Jun;97(6):2059-67. doi: 10.1210/jc.2011-3180. Epub 2012 Apr 3. PMID 22472563
- [Background] Wallace WH, Smith AG, Kelsey TW, Edgar AE, Anderson RA. Fertility preservation for girls and young women with cancer: population-based validation of criteria for ovarian tissue cryopreservation. Lancet Oncol. 2014 Sep;15(10):1129-36. doi: 10.1016/S1470-2045(14)70334-1. Epub 2014 Aug 14. PMID 25130994
- [Background] Demeestere I, Simon P, Dedeken L, Moffa F, Tsepelidis S, Brachet C, Delbaere A, Devreker F, Ferster A. Live birth after autograft of ovarian tissue cryopreserved during childhood. Hum Reprod. 2015 Sep;30(9):2107-9. doi: 10.1093/humrep/dev128. Epub 2015 Jun 9. PMID 26062556
- [Background] Imbert R, Moffa F, Tsepelidis S, Simon P, Delbaere A, Devreker F, Dechene J, Ferster A, Veys I, Fastrez M, Englert Y, Demeestere I. Safety and usefulness of cryopreservation of ovarian tissue to preserve fertility: a 12-year retrospective analysis. Hum Reprod. 2014 Sep;29(9):1931-40. doi: 10.1093/humrep/deu158. Epub 2014 Jun 22. PMID 24958067